CLINICAL TRIAL: NCT00888056
Title: Effect of Deep Brain Stimulation of the Hypothalamus/ Fornix on Memory Impairment in Patients With Alzheimer's Disease
Brief Title: Chronic Electrical Stimulation of Hypothalamus/Fornix in Alzheimer's Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-PP-01
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2009-04

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ARM A (Experimental): Bilateral chronic electrical stimulation of the hypothalamus/fornix
  Interventions: Procedure: Bilateral chronic electrical stimulation of the hypothalamus/fornix

INTERVENTIONS:
Procedure: Bilateral chronic electrical stimulation of the hypothalamus/fornix — Clinical, neuro-psychological, biological and imaging assessment will be performed 3 and one month before and 3, 6, 12 and 24 months after surgery. Bilateral electrodes (Medtronic 3389) will be implanted, under local anesthesia, by MR-guided frame-based stereotaxy, in the hypothalamic part of the fornix, before its entry in the mamillary body (well defined on T2 weighted sequences). Intra-operative stimulation will be used to search adverse effects or acute effects. Electrodes will be connected to the generator (Kinetra, Medtronic) under general anesthesia. Chronic high-frequency stimulation will be delivered immediately after surgery.

SUMMARY:
Alzheimer's Disease (AD) is the most common cause of dementia for which no treatment has shown consistent efficacy to stop or slow down the disease. Recent report of enhancement of memory abilities by bilateral chronic deep brain stimulation (DBS) of the fornix in the hypothalamus suggests that neuromodulation of circuits involved in memory processes may have therapeutic implications in AD patients with memory decline.

The primary objectives of this prospective, non-controlled, pilot study are to evaluate the feasibility and safety of DBS in AD patients with mild cognitive and memory impairment, and to evaluate the efficacy of DBS to slow down or stabilize this decline. Five patients with AD (DSM IV) diagnosed less than two years, with mild cognitive decline (MMSE 20-24), and specific impairment of episodic memory will be included in a 2-year period. The evaluation criteria for feasibility will be the proportion of patients undergoing the procedure, chronic stimulation and evaluation process without adverse event (AE). Efficacy will be evaluated using numerous cognitive and memory testing. Changes in behavioral and mood scales, and changes in hypothalamic functions (clinical, biological and hormonal assessment) will evaluate safety and tolerance. Clinical, neuro-psychological, biological and imaging assessment will be performed 3 and one month before and 3, 6, 12 and 24 months after surgery. Bilateral electrodes (Medtronic 3389) will be implanted, by MR-guided frame-based stereotaxy, in the hypothalamic part of the fornix, and then connected to the generator (Kinetra, Medtronic). Chronic high-frequency stimulation will be delivered immediately after surgery.

The investigators expect to slow down, or to stabilize the spontaneous decline of MMSE and ADAS scores after 6, 12 and 24 months of stimulation. In case of efficacy, DBS might offer to AD patient the possibility to slow down/stabilize their symptoms, which no other treatment can currently offer, and to increase their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* patients with AD (DSM IV) diagnosed less than 2 years
* age between 50 and 65
* mild cognitive decline (MMSE between 20 and 24)
* specific impairment of episodic memory (evaluated by Grober&Buschke scale)
* able to give and sign an informed consent
* affiliated to the French national health and pensions organization

Exclusion Criteria:

* associated DSM I axis pathology
* contra-indication to surgery or MRI
* preoperative MRI abnormalities
* retraction of consent by the patient
* decision of the promoter to stop the study

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2009-06

PRIMARY OUTCOMES:
Evaluation criteria for feasibility will be the proportion of patients undergoing the procedure, chronic stimulation and evaluation process without adverse event. | once time

SECONDARY OUTCOMES:
Efficacy will be evaluated using numerous cognitive and memory testing. Neuro-imaging changes after stimulation will be evaluate by morphological MRI and functional imaging (PET). Changes in behavioral and mood scales: evaluate safety | M-3, D-7, D7, M3, M6, M12, M24

CONTACTS AND LOCATIONS:
Overall Officials: Fontaine Denys, PhD, Principal Investigator — CHU de Nice - Service de Neurochirurgie - Hôpital Pasteur - 30 av de la voie Romaine - 06 100 Nice; ROBERT Philippe, PhD, Principal Investigator — CHU de Nice - CM2R - Hôpital de cimiez- 4 av reine Victoria 06001 Nice
Locations (1):
- CHU de Nice - 4 avenue Reine Victoria - Hôpital de Cimiez, Nice, Alpes-Maritimes, France